CLINICAL TRIAL: NCT00442533
Title: High Dose Indium-111 Pentetreotide Therapy in Somatostatin Receptor Expressing Neuroendocrine Neoplasms.
Brief Title: Safety and Efficacy Study of In-111 Pentetreotide to Treat Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radio Isotope Therapy of America (Other)
Collaborators: Excel Diagnostic Imaging Clinics (Unknown); Radiomedix, Inc. (Industry); CHI St. Luke's Health, Texas (Other)
Responsible Party: Principal Investigator, Ebrahim Delpassand, President and CEO, Radio Isotope Therapy of America
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-2247
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Neuroendocrine Tumors
Keywords: Carcinoid; Islet Cell Cancer; Paraganglioma; Pheochromocytoma
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Somatostatinoma; Paraganglioma; Pheochromocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indium-111 pentetreotide (Experimental): 4 cycles of 500 mCi treatments every 10-12 weeks
  Interventions: Drug: Indium-111 pentetreotide

INTERVENTIONS:
Drug: Indium-111 pentetreotide — 4 cycles of 500 mCi treatments every 10-12 weeks
  Other Names: NeuroendoMedix

SUMMARY:
The purpose of this study is to determine if High-dose 111In-Pentetreotide known as NeuroendoMedix®, is an effective treatment for Neuroendocrine Tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received first line standard chemotherapy and/or radiation therapy for neuroendocrine malignancy in the past and failed the therapy.
* Patients must have evidence of residual multifocal active tumor.
* All patients must sign an informed consent indicating the awareness of the investigational nature of the studies involved.
* All patients must have a Karnofsky performance status of at least 60.
* Patients must be greater than 18 years of age.
* Patients must have measurable and/or followable disease based on either clinical or radiologic exam.
* Sensitivity to Indium-111 pentetreotide or any of its components is an absolute contraindication to participation in this trial.
* An absolute contraindication is pregnancy as evidenced by the clinical condition, a positive pregnancy test (Beta type Human chorionic gonadotropin (β-HCG) or pelvic ultrasound).
* If patients have received prior radionuclide therapy of the same product, there must be documented response to that therapy and/or residual active stable disease.

Exclusion Criteria:

* Karnofsky performance status of 50 or less.
* Patients who are unable to give informed consent.
* Patients under 18 years of age. There will be no upper age discrimination.
* Patients who are pregnant or those potentially pregnant subjects not willing to practice effective contraceptive techniques during the study period.
* Patients with renal insufficiency as defined by a calculated creatinine clearance (based on age, weight and serum creatinine) of 39.9 ml/min or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2005-08; Primary Completion 2014-08-30 (Actual); Study Completion 2015-12-28 (Actual)

PRIMARY OUTCOMES:
Change in solid tumor dimensions by CT scan. | Baseline to post treatment CT scan performed 2-4 days after each cycle and 12and 24 weeks after treatments
  Change in diameters of measurable lesions on CT using RECIST. and will be classified into 4 groups.
  1. Complete response
  2. Partial response
  3. No change or stable disease
  4. Progression

SECONDARY OUTCOMES:
Frequency and severity of adverse events | up to 6 months following the last cycle of therap
  Frequency and severity of adverse events. All adverse events will be graded using NCI common toxicities criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim Delpassand, M.D., Principal Investigator — RITA Foundation
Locations (2):
- United States (2):
  - Excel Diagnostic Imaging Clinics, Houston, Texas
  - St. Lukes Episcopal Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided